CLINICAL TRIAL: NCT00175188
Title: A Roentgen Stereophotogrammetric Analysis and DEXA Study on Migration of Proximal Interphalangeal Joint Prostheses of the Hand. A Randomised Prospective Study of Cemented Versus Non-cemented Implants
Brief Title: An RSA and DEXA Study on Migration of Proximal Interphalangeal (PIP) Joint Prostheses of the Hand
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Zimmer Biomet (Industry); Avanta (Industry)
Responsible Party: Professor Kjeld Soballe, Aarhus University Hospital, Tage-Hansens Gade 2, 8000 Aarhus C
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20030240
Record Dates: First submitted 2005-09-10; First posted 2005-09-15 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-10

CONDITIONS: Osteoarthritis
Keywords: RSA; DEXA; Osteoarthritis; Finger implant; Micromotion; Bone density; Cement
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cemented PIP implant (Active Comparator): Avanta PIP
  Interventions: Device: Avanta (PIP joint implant with a titanium porous coating)
- Uncemented PIP implant (Active Comparator): Avanta PIP
  Interventions: Device: Avanta (PIP joint implant with a titanium porous coating)

INTERVENTIONS:
Device: Avanta (PIP joint implant with a titanium porous coating) — Implant is inserted at the time of surgery, after written consent
  Other Names: Avanta PIP implant, plasma-spray titanium coated

SUMMARY:
The purpose of this study is to compare the early migration and the periprosthetic bone changes of cemented versus non-cemented interphalangeal implants using Roentgen stereophotogrammetric analysis and dual energy x-ray absorptiometry (DEXA). Furthermore, a thorough occupational therapist evaluation on the functional progress prior to and after surgery will be assessed.

DETAILED DESCRIPTION:
There is a large patient group with primary osteoarthritis (OA) and secondary osteoarthritis due to joint-associated fractures, repeated trauma to the joint and surroundings, congenital joint-deformity, hyper mobility and diabetes. There are 2 preservative surgical treatment alternatives for PIP joint OA; namely arthrodesis and arthroplasty. Arthroplasty is the choice of treatment, when preserving motion is feasible, but patients can have excellent results with arthrodesis. There are several arthroplasty techniques including fibrous interposition, palmar plate advancement, metallic or metalloplastic hinges or one piece polymeric plastic hinge devices.

In this study, we use a 2 part metallic implant designed to minimize bone removal and preserve the collateral ligaments of the PIP joint providing a more stable joint particularly to imposed lateral forces. Preservation of the capsule with this prosthesis allows diversion of some of the transverse forces and axial torques from the prosthesis endosteal interface to the lateral cortices through the collateral ligaments. The semi-constrained design provides a more physiological articulation, and besides this the centered anatomical configuration allows a more reliable restoration of tendon movements to the joint. All of this probably diminishes the mechanical contribution to osteolysis and subsidence at the bone prosthesis interface and prolongs the time of survival of the prosthesis. All of these improvements on prosthetic design are very important and provide a better possibility for the patient to regain near-normal joint conditions.

The prosthesis has two components - one proximal and one distal. The proximal part has a symmetric shallow bicondylar anatomic configuration fixed on a stem for the intramedullary cavity of the proximal phalanx. The distal component is fabricated from polyethylene press-molded on a metal backing with a stem for the intramedullary cavity of the middle phalanx. Both implant parts are CoCr alloy with a coating of plasma sprayed porous titanium. Studies have shown that bone grows well into the titanium surface of experimental implants, but it is also fixed into bone using cement.

With the new type of PIP prostheses there is often excellent if not total long-term pain relief and little or no loss of movement. The stability becomes considerably better compared with older types of prostheses. The outcome is however dependant on the skill and experience of the surgeon.

The purpose of this study is to compare the early migration and the periprosthetic bone changes of cemented versus non-cemented interphalangeal implants. Furthermore a thorough occupational therapist evaluation on the functional progress prior to and after surgery will be assessed.

To evaluate both the implant-bone micromotions, metal markers have been placed on the implant preoperatively and other markers will be fixed in the phalangeal bone intra-operatively. This allows us to evaluate the implant micromotion with stereo x-rays by photogrammetric computer analyses called RSA at the Orthopaedic Center, Aarhus University Hospital. Follow-up stereo x-rays will be scheduled for 1 week, 6 weeks, 12 weeks, 6 months, 1 year and 2 years post-surgery. Periprosthetic bone density will be evaluated at 1 week, 1 year and 2 years upon inclusion at the Orthopaedic Center, Aarhus University Hospital. An occupational therapist will evaluate the joint range of motion, pain, edema and grip strength prior to surgery and throughout the 2 year follow up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with osteoarthrosis of the PIP joints.
* Patients with sufficient bone quality for implantation of a non-cemented prosthesis. This is estimated by the surgeon preoperatively.
* Informed written patient consent.
* Patients must read and understand Danish.

Exclusion Criteria:

* Patients with neuromuscular or vascular diseases in the affected upper extremity.
* Patients who, preoperatively, are found to have unsuitable bone quality for un-cemented arthroplasty fixation, for instance bone cysts not visible on x-ray.
* Patients who cannot refrain from taking non-steroidal anti-inflammatory drugs (NSAIDs) postoperatively including cox-2 inhibitors.
* Patients with previously diagnosed osteoporosis.
* Women who are pregnant or are at risk of getting pregnant during the time of investigation.
* Patients with rheumatoid arthritis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-06; Primary Completion 2010-08 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
PIP implant migration evaluated by RSA | 2010
Periprosthetic bone changes evaluated by DEXA | 2010

SECONDARY OUTCOMES:
Changes in pain, grip strength, edema and range of motion | 2010

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Søballe, MD, Prof., Principal Investigator — Orthopaedic Center, Aarhus University Hospital
Locations (1):
- Orthopaedic Center, Aarhus University Hospital, Aarhus, Denmark